CLINICAL TRIAL: NCT03485456
Title: Pharmacokinetic Evaluation and Tolerability of Dry Powder Tobramycin Via the Cyclops® in Children With Cystic Fibrosis
Brief Title: DPI-Tobra-Kind Cyclops® in Children With Cystic Fibrosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Onno Akkerman, Dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPI-Tobra-Kind
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Cystic Fibrosis
Keywords: Dry powder inhalation; Tobramycin
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tobramycin (Experimental): Tobramycin dry powder inhalation with 30, 60 and 90 mg. Nebulisation with 300 mg tobramycin
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: Tobramycin — Tobramycin dry powder inhalation with 30, 60 and 90 mg. Nebulisation with 300 mg tobramycin
  Other Names: Tobramycin dry powder

SUMMARY:
The goal is to investigate the pharmacokinetic properties of dry powder tobramycin via the Cyclops® at different dosages in children with cystic fibrosis, together with the local tolerability.

DETAILED DESCRIPTION:
Rationale: Cystic fibrosis is the most common life-shortening autosomal recessive disease among Caucasian populations. It is a chronic progressive disease causing deterioration of pulmonary function, and of general condition as well. Although it is a multisystem disease, the primary cause of death is respiratory failure, resulting from chronic pulmonary infection.

Pseudomonas aeruginosa is the predominant pathogen. The presence of P. aeruginosa in patients with CF is an unfavourable prognostic indicator and is associated with accelerated lung tissue destruction and loss of lung function, subsequently leading tot increased morbidity and mortality. Preventing, limiting and treating chronic infection with P. aeruginosa is therefore crucial in the management of CF, to improve survival and quality of life.

Currently most children with CF who are colonized with P. aeruginosa receive inhaled tobramycin every other month, mostly by use of a nebulizer. This delivery system however has several disadvantages. For example, the nebulisation itself and the cleaning of the nebulizer is time consuming. This places a high burden on a CF patient, especially for children, which will negatively influence compliance and quality of inhalation, thereby jeopardizing effective treatment. Therapy with a (disposable) dry powder inhaler (DPI) is less time consuming. Besides this, nebulisation brings the risk of auto-re-infection of the patient (contamination of nebulisation fluid and/or device). Other more technical disadvantages of nebulisation are a low lung deposition and pollution with tobramycin in the surrounding environment. With an efficient DPI, a three to six fold higher lung deposition compared to a nebulizer can be obtained. Nebulised tobramycin is used most in routine care, but sometimes a DPI is used, for example the Podhaler®. Although the dispersion behaviour of these dry powder systems is often good, the engineering processes make the products expensive, and the high excipient fractions make the inhaled powder doses high. Furthermore because these devices are not disposable, there is a risk of bacterial resistance development in the device. Next to this is the hygroscopic nature of tobramycin a risk for good dispersion when a used DPI is store inappropriately. In this situation powder residues in the inhaler become sticky or even liquefied when they absorb moisture from the air. There is one disposable DPI for tobramycin available, called the Cyclops®, but this DPI is not registered for children with CF yet. The investigators will therefore investigate dry powder tobramycin (DP tobramycin) in the Cyclops® in children with CF.

Objective: The main objectives are to investigate the pharmacokinetic properties of DP tobramycin via the Cyclops® at different dosages in children with CF, together with the local tolerability.

Study design: Single center, single ascending, single dose study.

Study population: 10 patients with CF, age 6 - 18 years.

Main study parameters/endpoints: The following pharmacokinetic parameters will be calculated: actual dose (dose minus remainder in inhaler after inhalation), AUC0-12 (area under the curve from 0 - 12 h), Cmax (maximum plasma concentration), Tmax (time to maximum plasma concentration), Ka (absorption rate constant), T1/2 el (terminal elimination half-life), CL/F (clearance following pulmonary administration (F= bioavailability)). Local tolerability of DP Tobramycin is determined by scoring adverse events, specifically coughing, and lung function measurement.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Target population of this study consists of children aged 6-18 years, because no information is available for inhalation of tobramycin using the Cyclops® in this population. Moreover, especially for children with CF a more easy to use and less time consuming treatment may improve their quality of life. Children participating in this study will receive instructions before using the DPI and their inspiratory flow will be tested. After each test dose serum samples will be collected with dry blood spot via a finger prick. To investigate safety, lung function tests will be performed before and 15, 30 and 90 minutes after inhalation and the occurrence of adverse events will be scored. Tobramycin is a registered drug for the treatment of chronic P. aeruginosa infection in CFpatients of 6 years and older. Inhalation of tobramycin is proven to be effective and safe in multiple studies. Dry powder tobramycin inhalation via the Cyclops® has been evaluated in adults with non-CF bronchiectasis. In this study a good drug dose - serum concentration correlation was obtained in adults, and the dry powder tobramycin inhalation via the Cyclops has been found safe with only mild tobramycin-related cough was reported once.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of CF and a positive sweat test or two CF-related mutations;
* Age 6 - 18 years
* Ability to breathe through a mouthpiece and to use the Cyclops
* Ability to perform pulmonary function tests
* Written informed consent (child and parents)

Exclusion criteria:

* Acute exacerbation of pulmonary infection
* FEV1 < 60%
* Subjects with known or suspected renal, auditory, vestibular of neuromuscular dysfunction, or with severe, active haemoptysis
* History of adverse events on previous tobramycin or other aminoglycoside use
* No concurrent use of cisplatin, cyclosporine, amphotericin B, cephalosporins, polymyxins, vancomycin and NSAID's

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
AUC 0-12 | 0-12 hours after dry powder inhalation
  Area under the curve from 0 - 12 h

SECONDARY OUTCOMES:
Cmax | 0-12 hours after dry powder inhalation
  maximum plasma concentration
Tmax | 0-12 hours after dry powder inhalation
  Time to maximum plasma concentration
Ka | 0-12 hours after dry powder inhalation
  Absorption rate constant
T 1/2 el | 0-12 hours after dry powder inhalation
  Terminal elimination half-life
CL/F | 0-12 hours after dry powder inhalation
  Clearance following pulmonary administration
Local tolerability | Before and 15, 30 and 90 minutes after inhalation
  Local tolerability determined by scoring adverse events, specifically coughing, and lung function

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Koppelman, Prof., Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No